CLINICAL TRIAL: NCT02150200
Title: Randomised Study Comparing Discharge 3 Days After Surgery to Home Within 24 Hours After Laparoscopic Hysterectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5717
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Women Who Undergo a Laparoscopic Hysterectomy for Benign Disease.
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A group : Conventional hospitalization (Other): Patients discharged after 3 days hospital stay after laparoscopic hysterectomy
  Interventions: Other: questionnaires
- B group : shorter stay (Experimental): Patients going home within 24 hours discharged the first day after laparoscopic hysterectomy.
  Interventions: Other: shorter hospitalization stay; Other: questionnaires

INTERVENTIONS:
Other: shorter hospitalization stay
  Arms: B group : shorter stay
Other: questionnaires

SUMMARY:
Hysterectomy is one of the most performed surgery in gynecologic surgery. Actually, 70 000 hysterectomies are performed each year in France. Laparoscopic surgery is in progression. The percentage of hysterectomies performed laparoscopically is increasing. The advantage of laparoscopy include fewer infections, less operative pain, faster recovery time and shorter hospital stay. In France, the average of hospital stay after laparoscopic hysterectomy reduced to 3-4 days.

The study hypothesis is that a shorter postoperative stay does not decrease the quality of life of the patients.

This study will compare the evolution of quality of life (with a questionnaire concerning measuring health related quality of life the Euroqol EQ-5D) of patients discharged after 3 days hospital stay to patients discharged the first day after a laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion criteria:

* age between 35 and 70.
* affiliation to a social security system
* signed informed consent form
* disponibility of an responsible and valid accompanying person during 48 hours
* home situation, less than one hour to go to an adapted structure of care
* access to a phone

Exclusion criteria:

* comorbidity which will automatically increase the period of hospital stay
* contraindication in laparoscopy
* difficulty to understand the protocol
* no social security cover

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessed by the Euroqol EQ-5D | up to 30th days after the laparoscopic hysterectomy.
  Measure of quality of life with a questionnaire concerning health related quality of life (the Euroqol EQ-5D).The patients will complete the questionnaire at up to 30th days after the laparoscopic hysterectomy.

SECONDARY OUTCOMES:
Quality of life with assessed by the short SF-36 score (the 36 items Short Form Health Survey). in pre-operative time and 30 days after the hysterectomy. | In pre-operative time and 30 days after the hysterectomy.
Patient satisfaction | Patient satisfaction assessed one month after intervention
Evaluation of pain by Visual Analog Scale for Pain and by analgesic drugs consumption | the day of intervention, 1 day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days and 30 days after intervention
Anxiety assessment by the State trait anxiety inventory forme Y-A | before intervention, the firt day, the second day, the third day after intervention, one week after intervention and one month after intervention.
Patient recovery and discharge after intervention assessed by Post-Anaesthetic Discharge Scoring System (PADSS score). | 8 hours after laparoscopic surgery
Comparison between a hospital stay of 3-4 days after laparoscopic hysterectomy costs and hospital stay of 1day after laparoscopic hysterectomy costs from the day of intervention until one month after intervention. | each day from the date of intervention untill one month after intervention.
  The assessment will take into account any case of rehospitalization
Perioperative morbidity | from intervention untill one month after intervention
Number of rehospitalization | one month after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hôptaux Universitaires de Strasbourg, Département de Gynécologie-Obstétrique, Strasbourg, France